CLINICAL TRIAL: NCT07016074
Title: Inorganic Nitrate (NaNO3) Prevention of Contrast-Associated Acute Kidney Injury
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Hitinder Gurm, Professor of Cardiovascular Medicine, Professor of Internal Medicine, and Chief Medical Officer, Medical School, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HUM00263577
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Kidney Injury, Acute
Keywords: Sodium Nitrate
MeSH Terms: conditions — Acute Kidney Injury | interventions — sodium nitrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Dispensing, and Labeling: The University of Michigan Research Pharmacy will compound sodium nitrate and placebo capsules. Placebo capsules will be compounded by filling a matching capsule with lactose.
  Interventions: Drug: Placebo
- Sodium Nitrate (Experimental): Dispensing, and Labeling: The University of Michigan Research Pharmacy will compound sodium nitrate and placebo capsules. Sodium nitrate powder will be measure and used for the active capsules with adding lactose as a filler.
  Interventions: Drug: Sodium Nitrate

INTERVENTIONS:
Drug: Sodium Nitrate — The study drug is sodium nitrate capsule at a dose of 12mmol of nitrate. This medication will be given orally 1-8 hours before the planned contrast administration and then once per day for a total of four doses.
  Other Names: Chili saltpeter
  Arms: Sodium Nitrate
Drug: Placebo — The placebo control medication will be a capsule filled with lactose that will be taken in the same manner and schedule as the sodium nitrate capsule
  Arms: Placebo

SUMMARY:
This pilot study is designed to test the logistics and recruitment of a trial testing the benefit of sodium nitrate in the prevention of contrast-associated kidney injury in a group of patients at high-risk.

ELIGIBILITY:
Inclusion Criteria:

* Planned coronary angiogram or contrast-enhanced CT scan.
* High-risk for contrast-associated acute kidney injury (AKI) with creatine/Glomerular filtration rate (GFR) within 90 days as defined as:

  1. Undergoing coronary angiogram with GFR <45 mL/min/1.73m2 OR
  2. Undergoing coronary angiogram with GFR <60 mL/min/1.73m2 and concurrent risk of AKI as defined by Hamilton et al. BMC2 risk prediction model ≥ 7%.

     OR
  3. Undergoing contrast-enhanced CT scan with GFR<45 mL/min/1.73m2
* If subject is a woman of child-bearing potential, subject agrees to the use of highly effective contraception starting at screening and during study participation.
* Ability to take oral medication and be willing to adhere to the study intervention regimen.
* Ability to understand and willingness to agree to an informed consent

Exclusion Criteria:

* Already fulfilling definition of acute kidney injury prior to contrast exposure by kidney disease improving global outcomes (KDIGO) criteria (absolute increase in creatinine from baseline of 0.3mg/dL or more OR relative increase in creatine of 50% or more from baseline).
* Primary indication for Percutaneous Coronary Intervention (PCI) including acute ST-segment elevation myocardial infarction
* End-stage renal disease actively on dialysis.
* Received any intravenous or intraarterial contrast within five days from planned contrast administration.
* Cardiac arrest within 14 days of planned contrast administration.
* Systolic blood pressure < 100mmHg or diastolic blood pressure <60mmHg OR currently receiving inotropes or vasopressors for hemodynamic support.
* History of hypersensitivity or known allergy to any of the components of the investigational product or placebo including sodium nitrate, inorganic nitrate, beet root juice, or lactose. This does not include lactose intolerance.
* Pregnancy or nursing female
* Participation in other investigational trials within the past 30 days prior to enrollment.
* Use of tadalafil within 48 hours, sildenafil or vardenafil within 24 hours, and avanafil within 12 hours of initiation of trial medication. If participant is on continuous dosing of tadalafil, sildenafil, vardenafil, or avanafil, they will be excluded from the trial. If participant is on intermittent dosing of tadalafil, sildenafil, vardenafil, or avanafil, patient agrees to withhold use of medication for duration of medication treatment extending 48 hours after the final dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Percent of participants receiving the first dose of blinded study drug within 1-8 hours prior to contrast exposure | Approximately 34 days
  Success is defined as greater than 80% of patients receiving the first dose of blind study drug within 1-8 hours prior to contrast exposure.
Percent of participants completing full course of 4 doses of blinded study drug | Approximately 34 days
  Success is defined as greater than 80% of patients completing the full course of 4 doses of blinded study drug
Percent of participants with 48-hour basic metabolic panel collected between 36-60 hours of contrast exposure | Approximately 34 days
  Success is defined as greater than 80% of patients having appropriately collected 48-hour basic metabolic panel collected 36-60 hours of contrast exposure
Percent of participants who had completion of clinical outcome monitoring at 30-day follow-up interview | Approximately 34 days
  Success is defined as greater than 80% of patients completing full clinical outcome monitoring at 30-day follow-up interview.
Percent of participants recruited to the trial for undergoing coronary angiogram | Approximately 34 days
  Success is defined as four or more patients being recruited into the study prior to coronary angiogram each month of the study averaged over the study period
Percent of participants recruited to the trial for undergoing a contrast-enhanced CT scan | Approximately 34 days
  Success is defined as four or more patients being recruited into the study prior to contrast-enhanced CT scan each month of the study averaged over the study period.

SECONDARY OUTCOMES:
Number of participants who develop of Contrast-Associated Acute Kidney Injury (CA-AKI) | Approximately 34 days
  As defined by creatinine measurement at 48 hours after contrast administration meeting Kidney Disease Improving Global Outcomes (KDIGO) criteria
Number of participants who had initiation of renal replacement therapy within 30 days of planned contrast administration for patients that did not have active need for dialysis prior to study enrollment | Approximately 34 days
Number of participants with all-cause mortality within 30 days of planned contrast administration as defined by cessation of life due to any cause | Approximately 34 days
Number of participants with major adverse cardiovascular events (MACE) | Approximately 34 days
  MACE is a composite endpoint of cardiovascular death, non-fatal myocardial infarction, and non-fatal stroke within 30 days of planned contrast administration
Number of participants with cardiovascular death within 30 days of planned contrast administration as defined by cessation of life deemed secondary to cardiovascular cause | Approximately 34 days
Number of participants with non-fatal myocardial infarction within 30 days of planned contrast administration | Approximately 34 days
Number of participants with non-fatal stroke within 30 days of planned contrast administration | Approximately 34 days
Number of participants with major adverse kidney events (MAKE) | Approximately 34 days
  MAKE is a composite outcome of death, new renal replacement therapy, or persistent renal dysfunction within 30 days of planned contrast administration. Persistent renal dysfunction is defined as creatinine value greater than or equal to 200% of baseline value at 30 days
Number of participants with persistent renal dysfunction at 30 days of planned contrast administration | Approximately 34 days
  Renal dysfunction is defined as creatinine value greater than or equal to 200% of baseline value at 30 days.
Number of participants with new onset hypotension | Approximately 34 days
Number of adverse events within 30 days of planned contrast administration | Approximately 34 days

CONTACTS AND LOCATIONS:
Overall Officials: Hitinder Gurm, MBBS, Study Chair — University of Michigan; David Hamilton, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No